CLINICAL TRIAL: NCT01677208
Title: A Randomized, Multi-center, Double-blind, Placebo-controlled Trial of Danhong Injection in the Treatment of Acute Ischemic Stroke
Brief Title: Danhong Injection in the Treatment of Acute Ischemic Stroke
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: China Food and Drug Administration (Other Government)
Responsible Party: Principal Investigator, Zhong Wang, Professor, China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DH20120423
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Acute Stroke
Keywords: Acute Ischemic Stroke; Randomized Controlled Trial; Traditional Chinese Medicine
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — danhong

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Danhong injection (Experimental): Based on the standard medical care, 40ml of Danhong injection, added into 250ml of 0.9% saline, given by continuous IV infusion at 2.5ml/min within 2 hours.
  Interventions: Drug: Danhong injection; Procedure: Standard medical care
- placebo (Placebo Comparator): Based on the standard medical care, 40ml of 0.9% saline as the placebo, added into 250ml of 0.9% saline, given by continuous IV infusion at 2.5ml/min within 2 hours.
  Interventions: Procedure: Standard medical care; Drug: placebo

INTERVENTIONS:
Drug: Danhong injection — A kind of injection made from two kind of Chinese herbs: Salvia miltiorrhiza and Safflower. 40ml Danhong injection added into 250ml 0.9% saline by an independent research nurse, sealed with brown bag in order to make the investigators and patients blinded, using brown infusion tube for infusion
  Arms: Danhong injection
Procedure: Standard medical care — Standard medical care is in accordance with China Guideline for the diagnosis and treatment of acute ischemic stroke (2010), including medical care for vital signs, control of temperature, blood pressure and glucose, improving cerebral blood circulation, antiplatelet treatment and nutritional supportive care.
Drug: placebo — 0.9% saline added into 250ml 0.9% saline by an independent research nurse, sealed with brown bag in order to make the investigators and patients blinded, using brown infusion tube for infusion.
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether Danhong injection is effective in the treatment of acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Female or male inpatients
* Age: 18 - 70 years.
* Clinical diagnosis of ischemic stroke causing a measurable neurological deficit defined as impairment of language, motor function, cognition and/or gaze, vision or neglect. Ischemic stroke is defined as an event characterized by the sudden onset of an acute focal neurologic deficit presumed to be due to cerebral ischemia after CT scan excludes hemorrhage.
* Clinical diagnosis of "Xueyu Zheng" (Blood Stasis Syndrome) as the scores of Chinese medicine symptoms scales of "Xueyu Zheng" in ischemic stroke ≥ 20. The Chinese medicine symptoms scales of "Xueyu Zheng" is defined as following (1)hemiplegia-10,(2)numbness of limbs-10，(3) dark face-9,(4)purple or dark lip-8,(5)Roughness of skin-4, (6) pain with fixed point-5, (7) purple or dark tongue-10,(8)ecchymosis on tongue-10,(9)purple sublingual vessel-10,(10)varicose sublingual vessel-8,(11)unsmooth pulse-8,(12)intermittent pulse-1.
* Onset of symptoms in 1 week prior to initiation of administration of study drug.
* Clinical diagnosis of cerebral anterior circulation obstruction.
* 4≤NIHSS<20.
* Patient is willing to participate voluntarily and to sign a written patient informed consent. Informed consent will be obtained from each patient or the subject's legally authorized representative or relatives, or deferred where applicable, according to the regulatory and legal requirements of the participating centers.

Exclusion Criteria:

* Evidence of intracranial hemorrhage (ICH) or other cerebral diseases (eg.vascular malformation, tumor, abscess or multiple sclerosis etc.)on the CT-or MRI-scan.
* Patients with thrombolysis or endovascular treatment.
* Known history of allergy or suspected allergic to the drug.
* Blood glucose 2.8 or > 16.8 mmol / l under the treatment of diabetes or with severe complications due to diabetes (eg. peripheral neuropathy, diabetic gangrene).
* Liver function impairment with the value of ALT or AST over 1.5-fold of normal value.
* Renal dysfunction with the value of serum creatinine over 1.5-fold of normal value.
* Severe cardiac dysfunction on echocardiogram or the grade of heart function over Ⅲ grade.
* History of prior stroke with mRS ≥2.
* Complicated with atrial fibrillation.
* Severe stroke as assessed by appropriate imaging techniques (eg. massive cerebral infarction including more than one lobe of brain or over 1/3 of blood-supply area of middle cerebral artery).
* Prior disable patients.
* Hemorrhagic tendency or recent severe or dangerous bleeding in 3 months.
* Suspected addicted into alcohol or drug abuse.
* With severe complications that would make the condition more complicated assessed by the investigator.
* Woman with pregnancy, lactation or positive result of pregnancy test, or women who want to be pregnant in recent 6 months.
* Woman who is under menstrual period.
* Patient who is participating in other trials or has been participated in other trials in recent 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1503 (Actual)
Dates: Start 2013-03-13 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale 0-1 (favourable outcome) at Day 90 | Day 90

SECONDARY OUTCOMES:
The Score of effect on symptoms of "Xueyue Zheng"(Blood Stasis syndrome) | Day 0, Day7, Day 14, Day 30, Day 60, Day 90
Barthel Index score ≥90 | Day 0, Day7, Day 14, Day 30, Day 60, Day 90
NIH stroke scale(NIHSS) | Day 0, Day7, Day 14, Day 30, Day 60, Day 90
  The improvement of the NIHSS score ≥4 or the NIHSS score of 0 to 1
EQ-5D scale | Day 0, Day 7, Day 14, Day 30, Day 60, Day 90
Global disability on mRS at Day 90. | Day 90
  The proportion of patients with mRS ≥3 at Day 90.
Incidence of new-onset major vascular events in 90 days | Day 90
  Major adverse vascular events include ischemic stroke, hemorrhagic stroke, TIA, myocardial infarction and vascular-related death.
Overall mortality at day 90 | Day 90
Incidence of severe hemorrhages in 90 days | Day 90
  The definition of "Severe hemorrhages" is in accordance with the GUSTO bleeding criteria, including fatal intracranial hemorrhage (ICH), symptomatic intracerebral hemorrhage (sICH) or which could result in substantial hemodynamic compromise requiring treatment.
Incidence of moderate hemorrhages in 90 days | Day 90
  The definition of "moderate hemorrhages" is in accordance with the GUSTO bleeding criteria, which requires blood transfusion but not results in hemodynamic compromise.
Documentation of adverse events (AEs) and serious AEs | 90 days

OTHER OUTCOMES:
The changes on the profiles of micro-RNA in 96 patients selected from certain centers | Day 0, Day 14, Day 90
The changes on the expression profiles of mRNA in 96 patients selected from certain centers | Day 0, Day 14, Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Wang, Professor, Principal Investigator — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences; Xing-quan Zhao, Professor, Principal Investigator — Beijing Tiantan Hospital; Yong-yan Wang, Professor, Study Chair — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences; Xiao-xi Du, Professor, Study Director — China Food and Drug Administration
Locations (62):
- China (62):
  - The Second Artillery General Hospital of Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Xinqiao Hospital of Third Military Medical University, Chongqing, Chongqing Municipality
  - Chongqing Three Gorges Central Hospital, Chongqing, Chongqing Municipality
  - Guangdong No.2 Provincial People's Hospital, Guangzhou, Guangdong
  - Guangzhou hospital of integrated Chinese and Western medicine, Guangzhou, Guangdong
  - The Second People's Hospital of Shenzhen, Shenzhen, Guangdong
  - The Second Central Hospital of Baoding City, Baoding, Hebei
  - Affiliated Hospital of Chengde Medical University, Chengde, Hebei
  - Handan Central Hospital, Handan, Hebei
  - The Second Affiliated Hopital of Harbin Medical University, Harbin, Helongjiang
  - The Second Chinese Medical Hospital of Luoyang City, Luoyang, Henan
  - Nanyang T.C.M. Hospital, Nanyang, Henan
  - Nanshi Hospital of Nanyang, Nanyang, Henan
  - The First Affiliated Hospital of Henan University of T.C.M., Zhengzhou, Henan
  - People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Zhengzhou NO.7 People's Hospital, Zhengzhou, Henan
  - Zhoukou Hospital of T.C.M., Zhoukou, Henan
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Zhongshan Hospital of Hubei Province, Wuhan, Hubei
  - Fifth Hospital in Wuhan, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Tianyou Hospital Affiliated to Wuhan University of Science & Technology, Wuhan, Hubei
  - Huangpi District Hospital of T.C.M., Wuhan, Hubei
  - Changsha Central Hospital, Changsha, Hunan
  - The First Hospital of Changsha, Changsha, Hunan
  - The second people's hospital of Hunan Province, Changsha, Hunan
  - Xiangya Hospital Central-south University, Changsha, Hunan
  - Nanjing Hospital of T.C.M., Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jilin Province People's Hospital, Changchun, Jilin
  - The Affiliated Hopital to Changchun University of Chinese Medicine, Changchun, Jilin
  - The First Hospital Affiliated to Jilin University, Changchun, Jilin
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Liaoyuan Traditional Chinese Medical Hospital, Liaoyuan, Jilin
  - Anshan Central Hospital, Anshan, Liaoning
  - Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning
  - Dandong First Hospital, Dandong, Liaoning
  - Panjin Central Hospital, Panjin, Liaoning
  - People's Liberation Army No.202 Hospital, Shenyang, Liaoning
  - The General Hospital of Shenyang Military, Shenyang, Liaoning
  - People's Liberation Army No.463 Hospital, Shenyang, Liaoning
  - Affiliated Hospital of Chifeng University, Chifeng, Neimenggu
  - Fenyang Hospital of Shanxi Province, Lüliang, Shanxi
  - The Second Affiliated Hospital to Shanxi Medical University, Taiyuan, Shanxi
  - Affiliated Hospital of Shanxi University of Chinese Medicine, Xianyang, Shanxi
  - The Second Affiliated Hospital of Shanxi University of T.C.M., Xianyang, Shanxi
  - Shanxi Province Hospital of T.C.M., Xi’an, Shanxi
  - The PLA Fourth Fifty-one Hospital, Xi’an, Shanxi
  - Shanxi Provincial People's Hospital, Xi’an, Shanxi
  - Teaching Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan
  - The First Affiliated Hopital of Chengdu Medical College, Chengdu, Sichuan
  - First Teaching Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality
  - Xin Hua Hospital of Zhejiang Province, Hangzhou, Zhejiang
  - Zhejiang Provincial Hospital of T.C.M., Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Huzhou Central Hospital, Huzhou, Zhejiang
  - Peking University First Hospital, Beijing
  - Tiantan Hospital Affiliated to Capital Medical University, Beijing
  - Xuan Wu Hospital Affiliated to Capital Medical University, Beijing

REFERENCES:
- [Derived] Li B, Wang Y, Lu J, Liu J, Yuan Y, Yu Y, Wang P, Zhao X, Wang Z. Evaluating the effects of Danhong injection in treatment of acute ischemic stroke: study protocol for a multicenter randomized controlled trial. Trials. 2015 Dec 9;16:561. doi: 10.1186/s13063-015-1076-4. PMID 26654631